CLINICAL TRIAL: NCT07139288
Title: Extracorporeal Shock Wave Versus Photobiomodulation Therapy for Chronic Ankle Instability
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Ramadan Ahmed, Assistant lecture, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P.T.REC/012/005760
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Chronic Ankle Instability, CAI
Keywords: extracorporeal shock wave, photobiomodulation, chronic ankle instability
MeSH Terms: interventions — Resistance Training; Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Inclusion criteria;
  The following criteria will be included:
  60 participants ranging in age from 18 to 65 years from both gender with a diagnosis of Chronic lateral ankle instability stage (II) (Schurz et al., 2023).
  Patients body mass index (BMI) are ranged from 18,5 to 25 (lee et al., 2022). The main presenting symptoms were ankle pain with restricted ROM that compromised activities of daily living (Schurz et al., 2023).
  All ankle sprains occurring more than four weeks before inclusion both recurrent sprain and CAI patients are included (Schurz et al., 2023).
  Mild to moderate severity of pain measured by NPRS scale (Srinivas, 2022). Partici¬pants had no history of ankle joint injuries or surgical procedures within the last year and injection treatment around the ankle joint within six months
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Exercise Program (Active Comparator): articipants receive a supervised therapeutic exercise program (strengthening, stretching, balance/proprioception). Standard care allowed.
  Interventions: Behavioral: therapeutic exercise program; Device: Extra corporeal shock wave therapy; Device: photobiomodulation Therapy
- ESWT (Experimental): participants will receive Extracorporeal Shock Wave Therapy (ESWT) in addition to standard care.
  Interventions: Device: Extra corporeal shock wave therapy
- Photobiomodulation (Experimental): Participants receive photobiomodulation therapy (low-level laser/LED) in addition to standard care.
  Interventions: Device: photobiomodulation Therapy

INTERVENTIONS:
Behavioral: therapeutic exercise program — Each subject completes four dynamic tasks, including ankle resistance exercises, resistance kinematic chain exercises, heel raise exercises, and BOSU ball exercises at 3 times per week for 4 weeks
  Other Names: balance and strength training
  Arms: Exercise Program
Device: Extra corporeal shock wave therapy — The extracorporeal shock waves will be delivered with 2,500 shockwave impulses (6 Hz), The intensity of extracorporeal shock waves is adjusted according to the patients' degree of tolerance to the pain. In the experimental group, the extracorporeal shockwave will apply to the anterior talofibular ligament, posterior talofibular ligament, calcaneofibular ligament, and tibialis anterior muscle.
  twice per week for 4 weeks
  Arms: ESWT; Exercise Program
Device: photobiomodulation Therapy — Photobiomodulation therapy will be performed with a laser an 810 nm wavelength, 0 ~ 500 mW adjustable and continuous power output, and a 0.4 cm beam diameter was used. The subjects in the group C will be treated with the laser at a dose of 239 J/cm2 (power: 100 mW; intensity: 796 mW/cm2; irradiation time: 5 min/point, 20 min in total) at 3 times per week for 4 weeks
  Other Names: PBM
  Arms: Exercise Program; Photobiomodulation

SUMMARY:
PURPOSE:

To Compare between the effect of extra corporeal shock wave and Photobiomodulation on pain level, ROM, muscle strength, function level, dynamic balance and thickness of ligament in patients with chronic ankle instability.

BACKGROUND:

Lateral ankle sprains are the most common lower limb musculoskeletal injury incurred by individuals who participate in sports and recreational physical activities Approximately 40% of individuals who sustain a LAS develop a condition known as chronic ankle instability (CAI) (Miklovic et al., 2018), The lateral ligamentous complex is the main structure affected in 80-85% of these injuries, which are originated from a sudden inversion or supination trauma (Mansur et al., 2021).

The ligament system plays a fundamental role in the ankle's stability and includes a talocrural complex and a subtalar complex that are functionally related. For the talocrural joint, three lateral collateral ligaments are present and one medial collateral ligament (Bonnel et al., 2010).

Physical examination is mostly the first diagnostic step in the assessment of ankle injuries. Imaging modalities such as ultrasonography (US) and magnetic resonance imaging (MRI) play a major role in providing a detailed depiction of ankle tendons and ligaments (Hosseinian et al., 2022).

The effect of ESWT is Higher multiplication of collagen fibers; faster organization of muscle fibers and vascularization by treatment with radial shockwaves (Schnurrer-Luke-Vrbanic et al., 2018), ESWT could improve pain, ankle instability, ankle function, dorsiflexion ROM, and dynamic balance in patients with CAI (Le et al., 2022).

Photobiomodulation Therapy (PBMT) is effective for patients with an ankle sprain. PBMT showed high effect size with a moderate level of evidence on pain intensity and is related to the PBMT intensity and frequency (Alayat et al., 2024).

HYPOTHESES:

There is no statistically significant effect of extra corporeal shock wave versus photobiomodulation on level of pain, ROM, muscle strength, function level, dynamic balance and thickness of ligament in patients with chronic ankle instability.

RESEARCH QUESTION:

Is there any effect of extra corporeal shock wave versus Photobiomodulation on pain level, ROM, muscle strength, function level, dynamic balance and thickness of ligament in patients with chronic ankle instability?

DETAILED DESCRIPTION:
The purpose of the study will be to investigate the effect of extracorporeal shock wave versus photobiomodulation therapy for chronic ankle instability Design of the study: A pre and posttest randomized controlled trial.

Subjects of the study:

participants will be chosen according to inclusive criteria. The sample size will be calculated depending on pilot study by power analysis (G power).

Group A: will receive exercise program include (Resistance Band Protocols, Resistance Kinematic Chain Exercises, Heel raise and Balance Exercise) at painful ankle.

Group B: as group A, plus the extra corporeal shock wave. Group C: as group A, plus the photobiomodulation

ELIGIBILITY:
Inclusion Criteria:

- 60 participants ranging in age from 18 to 65 years from both gender with a diagnosis of Chronic lateral ankle instability stage (II) (Schurz et al., 2023).

Patients body mass index (BMI) are ranged from 18,5 to 25 (lee et al., 2022). The main presenting symptoms were ankle pain with restricted ROM that compromised activities of daily living (Schurz et al., 2023).

All ankle sprains occurring more than four weeks before inclusion both recurrent sprain and CAI patients are included (Schurz et al., 2023).

Mild to moderate severity of pain measured by NPRS scale (Srinivas, 2022). no wounds in the ankle joint and calf (lee et al., 2022). Participants had no history of ankle joint injuries or surgical procedures within the last year and injection treatment around the ankle joint within six months (lee et al., 2022).

Exclusion Criteria:

* they had any medical condition that could cause ankle pain (arthritis, fracture, rheumatiod arthritis, any deformity of ankle and neurological condition).

Any individual who had previously suffered a musculoskeletal injury or surgery that could have influenced the measurement was also eliminated.

Any individual who had diagnosed a Chronic lateral ankle instability stage (I, III).

Acute foot trauma occurring from 7 days of injury (Srinivas, 2022).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-08-29 (Estimated); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Thickness of ligament in patients with chronic ankle instability. | Before and after treatment program for 1 month
  Thickness of ligaments (lateral ligaments) measure by sonography that done according to European Society of Musculoskeletal Radiology (ESSR) guidelines by an experienced radiologist
Function activity level | Before and after treatment program for 1 month
  The Arabic version of the IdFAI (IdFAI-Ar) questionnaire is effectively translated and cross-culturally adapted. It is valid, reliable, accurate, specific, and sensitive tool to determine ankle stability status. It obtained excellent reliability and strong validity to identify patients with FAI in both clinical practice and research

SECONDARY OUTCOMES:
pain assessment: | Before and after treatment program for 1 month
  The Numeric Pain Rating Scale measures the magnitude or intensity of pain or pain relief. The NPRS is an 11-point scale consisting of integers from 0 through 10; 0 representing ''no pain'' and 10 representing ''worst imaginable Pain
Ankle joint range of motion | Before and after treatment program for 1 month
  The ROM will be measured using baseline bubble inclinometer which has been shown to have high intra examiner reliability and validity ankle dorsiflexion, planterflexion, inversion and eversion will be measured with the participant in the supine position

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, EL Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Undecided